CLINICAL TRIAL: NCT01173510
Title: A Pilot Study to Determine if Raltegravir Eradicates HIV From Peripheral Blood Mononuclear Cells
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was not feasible due to facility budget and contractual issues.
Sponsor: Community Research Initiative of New England (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-184
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: HIV Infections; Acquired Immune Deficiency Syndrome
Keywords: HIV; AIDS; Atripla; Truvada; Raltegravir; Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome Virus
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir plus tenofovir/emtricitabine (Experimental)
  Interventions: Drug: Raltegravir plus Truvada
- Efavirenz/Emtricitabine/Tenofovir (Active Comparator)
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Raltegravir plus Truvada — Raltegravir 400 mg twice daily plus tenofovir/emtricitabine (Truvada) one tablet once daily
  Arms: Raltegravir plus tenofovir/emtricitabine
Drug: Atripla — Efavirenz/Emtricitabine/Tenofovir DF one tablet once daily
  Arms: Efavirenz/Emtricitabine/Tenofovir

SUMMARY:
Human Immunodeficiency Virus (HIV) infection is permanently established by integrating a deoxyribonucleic acid (DNA) copy into the human chromosome, a step also necessary to complete the Human Immunodeficiency Virus (HIV)replication cycle. Standard treatment of HIV infection suppresses Human Immunodeficiency Virus (HIV)replication and has not been able to eliminate Human Immunodeficiency Virus (HIV)from an infected person because of the integrated Human Immunodeficiency Virus (HIV). Raltegravir (RAL), the first approved antiretroviral (ARV) in a new class called integrase inhibitors, works by preventing integration of Human Immunodeficiency Virus (HIV). For participants with Human Immunodeficiency Virus (HIV)who have never taken antiretroviral medications, this research study will test whether Raltegravir (RAL), a recommended first-line ARV, can eliminate Human Immunodeficiency Virus (HIV)from key immune system cells.

DETAILED DESCRIPTION:
This is a phase IV study comparing RAL to EFV ability to clear the HIV from mononuclear cells. Participants will be randomized 2:1 to either RAL plus co-formulated FTC/TDF or EFV/FTC/TDF (Atripla). The study will last a minimum of 24 weeks. Participants will come in three days before the weeks 4 and 24 visits to receive a subcutaneous injection of G-CSF, an FDA-approved medication that mobilizes certain cells. A minimum of 5 visits will be required after baseline for blood draws, safety monitoring, or G-CSF injections.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects age 18 or older with HIV-1 infection
* CD4 cell counts greater than 200 cells/mm at screening
* Plasma HIV RNA > 1000 copies/mL
* Women of childbearing potential must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to eight weeks after the last dose of study drug. Women of childbearing potential includes any woman who has experienced menarche and who has not undergone successful surgical sterilization or who is not post-menopausal.

Exclusion Criteria:

* Previous exposure to antiretroviral medications used in the treatment of HIV-1 infection
* Evidence of genotypic or phenotypic resistance to most of the medications that will be used in the study (tenofovir, emtricitabine, and efavirenz) on a resistance assay obtained through the patient's primary care physicians as a standard of care test
* Women with a positive pregnancy test, who are pregnant, or who are breast feeding
* Sexually active non-sterilized men not using effective birth control if they have female partners who are of child-bearing potential
* Women of child-bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to eight weeks after the last dose of study drug
* Presence of any currently active AIDS-defining category C conditions according to the CDC Classification System for HIV Infection with the exception of stable cutaneous Kaposi's sarcoma
* Any active, clinically significant disease that in the opinion of the Principal Investigator may compromise the subject's safety during the trial
* Grade 3 or 4 Laboratory abnormalities as defined by a standardized grading scheme based on the DAIDS table - ACTG Toxicity Grading Scale elevations (except pre-existing diabetes mellitus with asymptomatic, non-fasting glucose grade 3 elevations, asymptomatic ≥ grade 3 fasting triglyceride or cholesterol elevations, and subjects with elevated indirect bilirubin)
* Active substance abuse or significant psychiatric illness that in the opinion of the Principal Investigator may interfere with study compliance
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness
* Known hypersensitivity to G-CSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-23 (Estimated); Primary Completion 2012-10-19 (Actual); Study Completion 2012-10-19 (Actual)

PRIMARY OUTCOMES:
Efficacy in eradicated HIV-1 integrated DNA from PBMCs | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating HIV-1 integrated DNA from peripheral blood mononuclear cells (PBMCs) in healthy HIV-infected participants who are naïve to antiretroviral therapy.
Efficacy in eradicating HIV-1 integrated DNA from CD34+ cells | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating HIV-1 integrated DNA from CD34+ cells mobilized from the bone marrow in healthy HIV-infected participants who are naïve to antiretroviral therapy.

SECONDARY OUTCOMES:
Efficacy in eradicating PBMC-associated early viral spliced mRNA | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating PBMC-associated early viral spliced mRNA (tat, rev, and nef) in healthy HIV-infected participants who are naïve to antiretroviral therapy.
Efficacy in eradicating PBMC-associated viral genomic RNA | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating PBMC-associated viral genomic RNA in healthy HIV-infected participants who are naïve to antiretroviral therapy.
Efficacy in eradicating CD34+-cell-associated early viral spliced mRNA | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating CD34+-cell-associated early viral spliced mRNA (tat, rev, and nef) in healthy HIV-infected participants who are naïve to antiretroviral therapy.
Efficacy in eradicating CD34+-cell-associated viral genomic RNA | 24 weeks
  To study the efficacy of Raltegravir plus Tenofovir DF/Emtricitabine versus Efavirenz/Emtricitabine/Tenofovir DF in eradicating CD34+cell-associated viral genomic RNA in healthy HIV-infected participants who are naïve to antiretroviral therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Clyde S Crumpacker, MD, Principal Investigator — Beth Israel Deaconess Medical Center - Division of Infectious Disease; Calvin J Cohen, MD, Principal Investigator — Community Research Initiative of New England

REFERENCES:
- See also: Community Research Initiative website — http://www.crine.org